CLINICAL TRIAL: NCT07224477
Title: A Phase 2, Randomized, Double-Blind, Comparator-Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of V540A in Healthy Females 16 to 26 Years of Age
Brief Title: A Clinical Study of V540A in Healthy Female Participants (V540A-005)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V540A-005; U1111-1314-2250 (Registry Identifier: UTN); 2024-518805-16-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2025-11-03; First posted 2025-11-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — Neu1 protein, mouse

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- V540A-2 (Experimental): Participants will receive vaccinations of V540A-2.
  Interventions: Biological: V540A-2
- V540A-3 (Experimental): Participants will receive vaccinations of V540A-3.
  Interventions: Biological: V540A-3
- GARDASIL®9 (Active Comparator): Participants will receive vaccinations of V503.
  Interventions: Biological: GARDASIL®9

INTERVENTIONS:
Biological: V540A-2 — Suspension administered via intramuscular (IM) injection.
  Arms: V540A-2
Biological: V540A-3 — Suspension administered via intramuscular (IM) injection.
  Arms: V540A-3
Biological: GARDASIL®9 — Suspension administered via IM injection.
  Other Names: G9; SILGARD®9; V503
  Arms: GARDASIL®9

SUMMARY:
Researchers are looking for new ways to prevent cancers related to human papillomavirus (HPV). HPV is a common virus that can cause an infection. There are many different types of HPV.

A standard vaccine to prevent HPV-related cancers is V503. V503 protects against 9 types of HPV. V540A is a study vaccine designed to protect against the same (shared) 9 HPV types plus other (unique) HPV types.

Researchers want to learn if V540A:

* Is safe and if people tolerate it
* Works as well as V503 to cause an immune response (the body's response to protect against infections and illnesses) to the shared HPV types.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Is in good health
* Has a lifetime history of 0 to 4 sexual partners of any sex/gender
* A participant assigned female sex at birth is eligible to participate if not breastfeeding during the study intervention period and for at least 30 days after the last dose of study intervention

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a history of severe allergic reaction (e.g., swelling of the mouth and throat, difficulty breathing, hypotension, or shock) that required medical intervention
* Has known or history of functional or anatomic asplenia
* Is currently immunocompromised or has been diagnosed as having congenital or acquired immunodeficiency, human immunodeficiency virus infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition
* Has thrombocytopenia or other coagulation disorder
* Has had a positive test for human papillomavirus (HPV)
* Has a history of recurrent respiratory papillomatosis or HPV-related head and neck cancer, or HPV-related anal lesions or anal cancer
* Has a history of an abnormal cervical biopsy result
* Has a history of HPV-related external genital lesions or external genital cancer, HPV-related vaginal lesions or vaginal cancer
* Has received a dose of any HPV vaccine before study entry
* Has received within 12 months before the Day 1 vaccination, is receiving, or plans to receive during the study, immunosuppressive therapies or other therapy known to interfere with the immune response
* Is currently receiving systemic steroid therapy or has received 2 or more courses of high-dose corticosteroids lasting at least 1 week in duration in the year prior to Day 1 vaccination
* Has received within the 3 months before the Day 1 vaccination, is receiving, or plans to receive during the study any immune globulin product

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 525 (Estimated)
Dates: Start 2026-07-20 (Estimated); Primary Completion 2028-04-04 (Estimated); Study Completion 2028-04-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience ≥1 Solicited Injection-site Adverse Event (AE) | Up to approximately 7 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs include redness (erythema), swelling (swelling), and pain or tenderness (pain). The number of participants who experienced at least 1 solicited injection-site AE from Day 1 through Day 5 post each vaccination will be reported.
Number of Participants Who Experience ≥1 Solicited Pyrexia AE | Up to approximately 7 months
  Pyrexia is defined as a temperature(s) ≥100.4°F (≥38.0°C). The number of participants with solicited pyrexia from Day 1 through Day 5 post each vaccination will be reported.
Number of Participants Who Experience ≥1 Vaccine-related Serious AE (SAE) | Up to approximately 7 months
  A vaccine-related SAE is any untoward medical consequence that results in death, is life-threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event which is determined by the investigator to be related to the vaccine. The number of participants who experienced at least 1 vaccine-related SAE will be reported.
Geometric Mean Titers (GMTs) to Each of the Shared Human Papillomavirus (HPV) Vaccine Types at Day 29 Postdose 3 | Up to approximately 7 months
  Antibodies to HPV types shared between V540A and GARDASIL®9 will be measured. Geometric mean titers of antibodies to HPV types at Day 29 postdose 3 will be reported.

SECONDARY OUTCOMES:
GMTs of Each of the Shared and Unique HPV Vaccine Types at Day 29 Postdose 1 | Up to 29 days
  Antibodies to HPV types shared between V540A and GARDASIL®9 and unique to V540A will be measured. Geometric mean titers of antibodies to HPV types at Day 29 postdose 1 will be reported.
GMTs of Each of the Shared and Unique HPV Vaccine Types at Day 29 Postdose 2 | Up to approximately 3 months
  Antibodies to HPV types shared between V540A and GARDASIL®9 and unique to V540A will be measured. Geometric mean titers of antibodies to HPV types at Day 29 postdose 2 will be reported.
GMTs to Each of the Shared and Unique HPV Vaccine Types at Day 29 Postdose 3 | Up to approximately 7 months
  Antibodies to HPV types shared between V540A and GARDASIL®9 and unique to V540A will be measured. Geometric mean titers of antibodies to HPV types at Day 29 postdose 3 will be reported.
Percentage of Participants with Seroconversion to Each of the Shared and Unique HPV Vaccine Types at Day 29 Postdose 1 | Up to approximately 2 months
  Seroconversion is defined as changing a participant's serostatus from seronegative at Day 1 to seropositive by Day 29 postdose 1. The percentage of participants with seroconversion to each of the shared and unique HPV vaccine types at Day 29 postdose 1 will be reported.
Percentage of Participants with Seroconversion to Each of the Shared and Unique HPV Vaccine Types at Day 29 Postdose 2 | Up to approximately 3 months
  Seroconversion is defined as changing a participant's serostatus from seronegative at Day 1 to seropositive by Day 29 postdose 2. The percentage of participants with seroconversion to each of the shared and unique HPV vaccine types at Day 29 postdose 2 will be reported.
Percentage of Participants with Seroconversion to Each of the Shared and Unique HPV Vaccine Types at Day 29 Postdose 3 | Up to approximately 7 months
  Seroconversion is defined as changing a participant's serostatus from seronegative at Day 1 to seropositive by Day 29 postdose 3. The percentage of participants with seroconversion to each of the shared and unique HPV vaccine types at Day 29 postdose 3 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com